CLINICAL TRIAL: NCT02420457
Title: Tracking Outcomes in Pain Patients Using Fitness Devices
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2949
Record Dates: First submitted 2015-03-31; First posted 2015-04-17 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Chronic Pain; Back Pain
Keywords: Fitness devices
MeSH Terms: conditions — Chronic Pain; Back Pain | interventions — Injections, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Back pain receiving epidural injection: Patients who have chronic back pain and are scheduled for an epidural injection to treat this pain will be receive a transforaminal epidural steroid injection as determined by routine care provider
  Interventions: Procedure: Epidural injection; Drug: Epidural steroid injection as determined by routine care provider

INTERVENTIONS:
Procedure: Epidural injection — After evaluation by their pain physician, if the clinician offers an epidural injection for their back pain, they will be followed for this study before and after the injection.
Drug: Epidural steroid injection as determined by routine care provider — Betamethasone Triamcinolone Dexamethasone Methylprednisolone Lidocaine Bupivacaine Ropivacaine Normal saline

SUMMARY:
The investigators are assessing the validity of fitness devices as surrogate measures of chronic pain survey outcomes.

DETAILED DESCRIPTION:
The investigators are attempting to validate the usage of personal fitness trackers against the classical survey tools used. These devices are known to be of use in measuring activity and sleep in healthy patients but their use in chronic pain patients has not been assessed. This study will follow participants with chronic back pain undergoing treatment to see if changes in clinical course can be captured with these fitness devices.

ELIGIBILITY:
Inclusion Criteria:

* Back pain which may benefit from epidural injection
* Assenting to epidural injection for back pain

Exclusion Criteria:

* Inability to wear fitness tracking device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic back pain
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-03; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Association of percent improvement in pain and number of steps. | Follow-up assessment approximately 2-4 weeks following epidural procedure.
  Linear regression will be used to determine the association of change in percent improvement of pain (assessed at baseline and follow-up) and number of steps taken on average the week of the assessment. Increased beta-coefficient from linear regression demonstrates that increased improvement in pain is related to an increased number of steps indicating improved mobility. If the beta coefficient from the linear regression is negative, this indicates that percent improvement in pain is associated with decreased number of steps and reduced mobility.

SECONDARY OUTCOMES:
Change in pain severity following procedure | Follow-up timepoint approximately 2-4 weeks following procedure
  Pain will be assessed by using a Visual Analog Scale (VAS) where scores range from 0 = no pain to 100 = worst possible pain. An increase in pain scores from baseline represent disease progression and decrease represent clinical response to treatment. VAS will be assessed prior to treatment and then at a followup assessment.
Association in minutes slept as measured by fitness device and percent improvement in pain | Follow-up assessment approximately 2-4 week following procedure
  Linear regression will be used to determine the association of change in percent improvement of pain (assessed at baseline and follow-up) and number of minutes slept on average the week of the assessment. Increased beta-coefficient from linear regression demonstrates that increased improvement in pain is related to an increased number of steps indicating improved mobility. If the beta coefficient from the linear regression is negative, this indicates that percent improvement in pain is associated with decreased number of steps and reduced mobility.
Change in survey measures of pain | Follow-up assessment approximately 2-4 weeks following the procedure.
  Conglomerate survey device of brief pain inventory, roland morris disability questionnaire, and oswestry disability index. The investigators will measure baseline survey data before the treatment and then at follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Mauck, MD PhD, Principal Investigator — Assistant Professor
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States